CLINICAL TRIAL: NCT04351282
Title: SBRT for Oligo-metastatic Lesions After Systemic Treatment of Primary Metastatic Nasopharyngeal Carcinoma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xiayun He, MD, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPC-SBRT
Record Dates: First submitted 2020-04-02; First posted 2020-04-17 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Nasopharyngeal Carcinoma; Metastasis; Stereotactic Body Radiation Therapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Neoplasm Metastasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SBRT (Experimental): 4-6 cycles of chemotherapy±immunotherapy and radical radiotherapy for nasopharyngeal tumors were given. SBRT for oligometastatic lesions will be assigned to those who got PR,SD after systemic treatment.
  Interventions: Radiation: SBRT

INTERVENTIONS:
Radiation: SBRT — SBRT for oligometastatic lesions will be assigned to those who got PR,SD after systemic treatment.

SUMMARY:
Primary metastatic NPC patients received chemotherapy± immunotherapy, radiation for primary tumors and SBRT for metastatic lesions.

DETAILED DESCRIPTION:
The eligible patients will receive 4-6 cycles chemotherapy±immunotherapy and radical radiotherapy for nasopharyngeal tumors. Then, SBRT for oligometastatic lesions will be assigned to eligible patients. The efficacy and side-effect will be evaluated and analyzed. The relation of liquid biopsy data with treatment outcome（such as EBV DNA, CTCs, CTC subtype，PD-L1 and so on）will be valued.

ELIGIBILITY:
Inclusion Criteria:

* Histologically conformed initial metastatic non-keratinizing nasopharyngeal carcinoma (according to the 8th edition of AJCC/UICC stage system) and no PD was observed in eligible patients after comprehensive treatment (chemotherapy±immunotherapy+radiotherapy to primary tumor). Then, the metastic lesions were PR/SD, and met the following requirement: the metastatic lesions ≤5 and metastatic organs ≤2, no more than 3 metastastic lesions for a single organ (diameter ≤ 5cm)
* age 18-70 years old
* Karnofsky scores ≥70
* Estimated life ≥ 6 months
* Adequate organ function including the following: Absolute neutrophil count (ANC) >= 2.0 * 109/l; Platelets count >= 100 * 109/l ;Hemoglobin >= 90 g/dl; Creatinine clearance >= 60 ml/min; For patients without liver metastasis, AST and ALT <= 1.5 times institutional upper limit of normal (ULN), Total bilirubin <= 1.5 times institutional ULN; For patients with liver metastasis, AST and ALT <= 3 times institutional upper limit of normal (ULN), Total bilirubin <= 3 times institutional ULN, with normal coagulation function, child-pugh grade A or B, normal liver tissue volume >700 mL
* Signed written informed consent

Exclusion Criteria:

* Patients who achieve complete remission after comprehensive treatment
* Pathology confirmed as second primary tumor
* Received radiotherapy at the corresponding site before, and overlapped with the site of this radiotherapy
* Femoral bone metastasis
* With serious medical complications and contraindications of radiotherapy
* With uncontrollable malignant pleural effusion
* Positive pregnancy test for women of childbearing age or lactating women
* Uncontrolled or active infections, such as immunodeficiency or HIV infection
* Active mental disorder or other mental disorder that affects the patient's ability to sign informed consent and understanding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | up to 3 years
  From date of diagnosis until the date of death from any cause

SECONDARY OUTCOMES:
Progress free survival | up to 3 years
  From date of diagnosis until the date of first documented progression or date of death from any cause, whichever came first
Previous Metastatic Progression Free Survival | up to 3 years
  From date of diagnosis until the date of first documented previous metastatic progression or date of death from any cause, whichever came first
New Metastatic Free Survival | up to 3 years
  From date of diagnosis until the date of first documented new metastasis
Adverse Event | up to 3 years
  Number of Participants with acute or late toxicities

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided